CLINICAL TRIAL: NCT04994288
Title: Efficacy and Safety of Once-weekly Supaglutide Versus Placebo in Patients With Type 2 Diabetes Suboptimally Controlled on Diet and Exercise: A Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: A Study of Efficacy and Safety of Supaglutide in Type 2 Diabetes Patients(SUPER-1)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Yinnuo Pharmaceutical Technology Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YN011-301
Record Dates: First submitted 2021-07-28; First posted 2021-08-06 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2023-08

CONDITIONS: Type2 Diabetes

STUDY DESIGN:
Intervention Model Description: This clinical trial includes dosage determination (Phase IIb) and efficacy confirmation stage(Phase III ).
  Subjects were randomly assigned to once-weekly subcutaneously injected Supaglutide 1mg, 2mg, 3mg and placebo according to a 2:2:2:1 ratio. During the IIb period, after Interim analysis and IDMC confirmed the RP3D high and low doses, subjects were randomly assigned to Supaglutide RP3D high dose, RP3D low dose and placebo group according to a 2:2:1 ratio.
Who Masked: Participant, Investigator
Masking Description: This includes a 24-week double-blind treatment period, followed by a 28-week open-label treatment period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supaglutide RP3D high dose (Experimental): during the IIb phase 140 subjects were randomly assigned to supaglutide 1mg, 2mg ,3mg and placebo ; when these subjects meets the 12wks HbA1C result, an interim analysis will be made andRP3D high dose is confirmed by IDMC accoding to interim analysis. So during the phase 3 , subjets will be assigned to RP3D hign dose, RP3D low dose and placebo
  Interventions: Biological: Supaglutide injection
- supaglutide RD3D Low dose (Experimental): during the IIb phase 140 subjects were randomly assigned to supaglutide 1mg, 2mg ,3mg and placebo ; when these subjects meets the 12wks HbA1C result, an interim analysis will be made and RP3D high dose is confirmed by IDMC accoding to interim analysis. So during the phase 3, subjets will be assigned to RP3D hign dose, RP3D low dose and placebo
  Interventions: Biological: Supaglutide injection
- placebo (Placebo Comparator): placebo injection
  Interventions: Other: placebo injection

INTERVENTIONS:
Biological: Supaglutide injection — Supaglutide 1mg/0.5ml , 2mg/0.5ml ,3mg /0.5ml
  Arms: Supaglutide RP3D high dose; supaglutide RD3D Low dose
Other: placebo injection — placebo injection 0.5ml
  Arms: placebo

SUMMARY:
This is a study to evaluate the efficacy and safety of Supaglutide injection in the treatment of type 2 diabetes patients with poor glycemic control after diet and exercise intervention.

This trial includes dosage determination (Phase IIb) and efficacy confirmation stage(Phase III).

The primary outcome of the phase IIb period is to preliminarily evaluate the efficacy and safety of Supaglutide and to provide the recommended dosage for the Phase 3 period after 12-week treatment.

The primary outcome of the Phase III period is to evaluate the efficacy and safety of Supaglutide after 24-week, double-blind treatment. The secondary outcome is to evaluate the efficacy and safety of Supaglutide after 24-week, double-blinded plus 28-week, open-label treatment period.

DETAILED DESCRIPTION:
This trial includes a 2-week screening period, a 4-week induction period, a 24-week double-blind treatment period and a 28-week open-label treatment period, followed by a 4-week follow-up period and a follow-up visit.

sample size was calculated to be 552, including 140 subjects in the period of Phase IIb and 412 subjects in the period of Phase III.

Subjects were randomly assigned to once-weekly subcutaneously injected Supaglutide 1mg, 2mg, 3mg and placebo according to a 2:2:2:1 ratio. During the IIb period, after Interim analysis and IDMC(Independent Data Monitoring Committee) confirmed the RP3D ( Recommended phase 3 dosage ) high and low doses, subjects were randomly assigned to Supaglutide RP3D high dose, RP3D low dose and placebo group according to a 2:2:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged from 18 to 75;
2. Type 2 diabetes diagonsed at least 8 weeks and has not received any glucose-lowering medication within 8 weeks prior to screening;
3. During screening, HbA1c: 7.5% ≤ HbA1c ≤ 11%;
4. Before randomization : 7.5% ≤ HbA1c ≤ 10.5%;
5. During screening and before randomization: FPG< 13.9 mmol/L
6. 18.5 kg/m2 ≤ BMI ≤ 35 kg/m2;
7. without birth plan and voluntarily take effective contraceptive measures;
8. fully understood the study, voluntarily entered the study and signed the informed consent.

Exclusion Criteria:

1. Diabetes other than Type 2;
2. Any DPP-4 inhibitors and / or GLP-1 analogues were used within 3 months before screening;
3. Continuous use of insulin for more than 14 days in the previous year;
4. C-Peptide <0.3 nmol/L;
5. Diabetic ketoacidosis, diabetic lactic acidosis or hyperosmolar non ketonic diabetic coma occurred within 6 months before screening;
6. Unstable proliferative retinopathy or macular lesion, severe diabetic neuropathy, intermittent claudication or diabetic foot occurred within 6 months before screening;
7. Severe hypoglycemia occurred within 6 months before screening
8. Severe trauma infection or operation within one month before screening;
9. Blood donation or massive blood loss or transfusion within 3 months ;
10. Suspected active infection ;
11. Growth hormone therapy was performed within 6 months before screening;
12. Patients having received corticosteroid continuous ≥ 7 days through within 2 months ;
13. use any drugs or surgery with weight control effect within 2 months;
14. weight change of more than 5% within 3 months;
15. mean systolic pressure (SBP) ≥ 160mmhg and / or DBP ≥ 90 mmHg at screening, or new/changed antihypertensive drugs or adjusted dosage of antihypertensive drugs within 4 weeks before screening or before induction period
16. with a history of severe cardiovascular disease, high risk of stroke/stroke within 6 months before screening;
17. with a history of acute or chronic pancreatitis, symptomatic gallbladder , pancreatic injury and other risk factors for pancreatitis, or with blood amylase and/or blood lipase ≥1.5 times the upper limit of normal (ULN) at the time of screening or before randomization;
18. Calcitonin level ≥50 ng/L (pg/mL) during screening;
19. with a history of medullary thyroid cancer, multiple endocrine neoplasm (Men) 2A or 2B syndrome, or related family history;
20. with clinically significant abnormal gastric emptying , severe chronic gastrointestinal diseases , long-term use of drugs that have a direct impact on gastrointestinal peristalsis , or having undergone gastrointestinal surgery within 6 months before screening, are not suitable to participate in this clinical study according to the evaluation of the researchers;
21. suffering from hematological diseases or any disease causing hemolysis or erythrocyte instability ;
22. Uncontrolled hyperthyroidism or hypothyroidism;
23. with hemoglobinopathy that may affect the determination of HbA1c levels;
24. HBsAg, HCV-Ab, HIV-Ab, TPAb or COVID-19 nucleic acid tested positive;
25. serious mental illness;
26. drinking more than 14 standard units weekly within 6 months before screening ;
27. a history of organ transplantation or other acquired or congenital immune system diseases;
28. allergic to the active ingredients (GLP-1 and GLP-1 analogues) of the study drug;
29. clear contraindications for the use of metformin;
30. Any of the following conditions: the pacemaker was installed when screened; no pacemaker was installed, but 12 lead ECG showed degree II or III atrioventricular block, long QT syndrome or QTc interval ≥ 450ms (fridericia formula was used to calculate QTCF); Patients with New York Heart Function Classification III or IV; Or other abnormal cardiac function with clinical significance that is not suitable for clinical research judged by researchers;
31. acute or chronic hepatitis, or whose laboratory examination indexes meet one of the following criteria at the time of screening or before randomization : alanine aminotransferase (ALT) level ≥ 2.5 fold ULN, aspartate aminotransferase (AST) ≥ 2.5 fold ULN, fasting triglyceride (TG) > 5.7 mmol/L or 500 mg/dl; the glomerular filtration rate (EGFR) < 60 ml/min/1.73 m2 was calculated by CKD-EPI (epi - (SCR)) formula;
32. participated in clinical trials of other drugs or devices within 3 months before screening;
33. Medication compliance in the lead-in period was < 75% or > 125%;
34. Any other situation that researchers think may affect the patients' informed consent or compliance with the trial protocol, or the patients' participation in the trial may affect the trial results or their own safety.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 547 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-08-16 (Actual)

PRIMARY OUTCOMES:
HbA1c | 12 weeks for phase IIb; 24weeks and 52 weeks for phase III
  The change in mean HbA1c concentrations (%)from baseline with Supaglutide versus placebo

SECONDARY OUTCOMES:
FPG | 12 weeks for phase IIb; 24weeks and 52 weeks for phase III
  Changes in FPG (mmol/L) relative to baseline
HbA1c<7.0% and <6.5% | 12 weeks for phase IIb; 24weeks and 52 weeks for phase III
  The proportion of participants who achieved HbA1c target (HbA1c<7.0% and <6.5% Patient percentage)
Fasting insulin | 12 weeks for phase IIb; 24weeks and 52 weeks for phase III
  Fasting insulin changes（pmol/L) relative to baseline
fasting C-peptide | 12 weeks for phase IIb; 24weeks and 52 weeks for phase III
  Fasting C-peptide changes (nmol/L) relative to baseline
fasting glucagon | 12 weeks for phase IIb; 24weeks and 52 weeks for phase III
  fasting glucagon changes (pg/ml) relative to baseline
Area under the curve of blood glucose | 12 weeks for phase IIb; 24weeks and 52 weeks for phase III
  Area under the curve of blood glucose(AUC0-120min,mmol/L) during the MMTT
Area under the curve of insulin | 12 weeks for phase IIb; 24weeks and 52 weeks for phase III
  Area under the curve of insulin (AUC0-120min,pmol/L) during the MMTT
Area under the curve of C-peptide | 12 weeks for phase IIb; 24weeks and 52 weeks for phase III
  Area under the curve of C-peptide (AUC0-120min,nmol/L) during the MMTT
fasting lipid profiles | 12 weeks for phase IIb; 24weeks and 52 weeks for phase III
  Changes in fasting lipid profiles relative to baseline(mmol/L)
weight | 12 weeks for phase IIb; 24weeks and 52 weeks for phase III
  Weight change from baseline(kg)
salvage treatment | 12 weeks for phase IIb; 24weeks and 52 weeks for phase III
  Percentage of subjects receiving salvage treatment(%)

CONTACTS AND LOCATIONS:
Overall Officials: Dalong Zhu, M.D,Ph.D, Principal Investigator — Nanjing trum tower hospital affiliated to Nanjing university school of medizine
Locations (1):
- Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu D, Ma J, Wang W, Shi B, Dong X, Bian F, Li Q, Wang Y, Jiang C, Wang X, Wang K, Ling H, Shi X, Cheng Z, Yuan G, Li L, Su X, Lu Y, Song W, Zhang Y, Hu W, Zhang X, Wang H, Liu Y, Li J, Zhang L, Liu Y, Sun X, Wang X, Zhang K, Zhao Y, Zhang L, Pan T, Li P, Li S, Zhou H, Jiang C, Zheng X, Ni L, Feng B, Li F, Piao L, Jin H, Liu Y, Cao H, Li Y, Cai H, Mao H, Liang Y, Guo J, Wang Y, Li Y, Xu N, Zhang J, Zhang Q, Pang W, Yu J, Xu Y, Zhou Y, Li Y, Wang Q. Efficacy and safety of efsubaglutide alfa in individuals with type 2 diabetes (SUPER1): a randomised, double-blind, placebo-controlled, Phase IIb/III trial. Diabetologia. 2025 Nov 21. doi: 10.1007/s00125-025-06593-2. Online ahead of print. PMID 41272211
- [Derived] Wang Q, Jiang F, Xu Y, Lei Y, Zhang L, Sun X. Exposure-Response Analysis of Efsubaglutide Alfa in Patients with Type 2 Diabetes Mellitus. Clin Pharmacokinet. 2025 Dec;64(12):1785-1797. doi: 10.1007/s40262-025-01570-9. Epub 2025 Oct 17. PMID 41107649
- [Derived] Lou YR, Xu YL, Xiong Y, Deng C, Wang Q. Population Pharmacokinetics of Efsubaglutide Alfa in Healthy Subjects and Subjects with Type 2 Diabetes. Clin Pharmacokinet. 2025 Apr;64(4):533-552. doi: 10.1007/s40262-025-01475-7. Epub 2025 Feb 17. PMID 39961992